CLINICAL TRIAL: NCT05863221
Title: A Phase IV, Open-Label, Randomized, Active-controlled, Single-Center Study of ZYNRELEF® for Postoperative Analgesia After Laparoscopic Sleeve Gastrectomy
Brief Title: ZYNRELEF® for Postoperative Analgesia After Laparoscopic Sleeve Gastrectomy
Acronym: HeronBariatric
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Yannis Raftopoulos (Other)
Collaborators: Heron Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Dr. Yannis Raftopoulos, Director of Weight Management Program, Holyoke Medical Center
Organization: Holyoke Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Heron Holyoke 1
Record Dates: First submitted 2023-05-09; First posted 2023-05-17 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain, Acute; Bariatric Surgery Candidate; Postoperative Pain
Keywords: Postoperative Pain; Bariatric Surgery; Opioid use
MeSH Terms: conditions — Pain, Postoperative | interventions — bupivacaine-meloxicam drug combination

STUDY DESIGN:
Intervention Model Description: This is a phase IV open-label, randomized, active-controlled study on subjects undergoing laparoscopic sleeve gastrectomy under general anesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): ZYNRELEF® up to 200 mg/ 6mg ( 7ml vial) via instillation at all incision sites in addition to 30 ml of 0.5% Ropivacaine + 10mg dexamethasone. Postoperatively, intermittent IV acetaminophen will be administered as per need till discharge.
  Interventions: Drug: ZYNRELEF 200Mg-6Mg Extended-Release Solution
- Group 2 (No Intervention): 30 ml of 0.5% Ropivacaine and 10mg dexamethasone into all surgical sites and intermittent IV acetaminophen as per need till discharge.

INTERVENTIONS:
Drug: ZYNRELEF 200Mg-6Mg Extended-Release Solution — ZYNRELEF® is an extended-release, fixed-ratio combination product that contains bupivacaine (a local anesthetic as the free base) and low-dose meloxicam (an NSAID) incorporated in a bioerodible polymer (termed Biochronomer®).
  Arms: Group 1

SUMMARY:
Approximately 120 subjects will be randomized into 1 of the following 2 treatment groups in a 1:1 ratio:

Group 1: ZYNRELEF® up to 200 mg/ 6mg ( 7ml vial) via instillation at all incision sites in addition to 30 ml of 0.5% Ropivacaine + 10mg dexamethasone. Postoperatively, intermittent IV acetaminophen will be administered as per need till discharge.

Group 2: 30 ml of 0.5% Ropivacaine and 10mg dexamethasone into all surgical sites and intermittent IV acetaminophen as per need till discharge.

Primary Objective:

To compare the efficacy and duration of analgesia achieved following the instillation of ZYNRELEF® all incision sites in addition to Ropivacaine with dexamethasone + postoperative IV acetaminophen, to the standard treatment of Ropivacaine with dexamethasone + postoperative IV acetaminophen in subjects undergoing laparoscopic sleeve gastrectomy.

Secondary Objectives:

1. To evaluate additional efficacy parameters, including opioid load, in this study population.
2. To determine the impact of ZYNRELEF® on the cost of pain management.
3. To assess the time taken to resume exercise after discharge.
4. To assess the adverse events reported following the use of ZYNRELEF®.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide written informed consent.
2. Is able to adhere to the study visit schedule and complete all study assessments.
3. Is male or female or other, and ≥18 years of age at screening.
4. Is scheduled to undergo laparoscopic sleeve gastrectomy under general anesthesia
5. Has an American Society of Anesthesiologists Physical Status of I, II, or III.
6. Female subjects are eligible only if all the following apply:

   * Not pregnant (female subjects of childbearing potential must have a negative urine pregnancy test at screening and on Day 1 before surgery).
   * Not lactating.
   * Not planning to become pregnant during the study.
   * Is surgically sterile (eg, has had a bilateral tubal ligation); or is at least 2 years postmenopausal; or is in a monogamous relationship with a partner who is surgically sterile; or is practicing abstinence or agrees to use double-barrier contraception in the event of sexual activity; or is using an insertable, injectable, transdermal, or combination oral contraceptive approved by applicable regulatory authorities for greater than 2 months prior to screening and commits to the use of an acceptable form of birth control for the duration of the study and for 30 days after study drug administration. Note: women in only a same-sex relationship do not need to meet this criterion.

Exclusion Criteria:

1. Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to Ropivacaine (or other local anesthetics), meloxicam, acetaminophen, ketamine, fentanyl, hydromorphone or dexamethasone. Subjects in all cohorts must not have any contraindications to any of the protocol-specified drugs (Ropivacaine, bupivacaine, lidocaine, meloxicam, fentanyl, ketamine, acetaminophen, hydromorphone or dexamethasone).
2. Has been administered Ropivacaine within 5 days prior to the scheduled surgery.
3. Has been administered any local anesthetic within 72 hours prior to the scheduled surgery, other than for pretreatment prior to a needle placement, to treat an AE that occurs after signing the ICF, or to decrease venous irritation (eg, caused by propofol, in which case no more than a single administration of lidocaine 1% 20 mg IV may be administered).
4. Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of the study drug (whichever is longer). Note that for purposes of this exclusion criterion, inhaled, ophthalmic, and over-the-counter steroids are not considered systemic.
5. Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments. Conditions may include but are not limited to, any of the following:

   1. History of asthma or urticarial/ allergic-type reactions after taking aspirin or NSAIDs.
   2. History of clinically significant cardiac abnormality such as myocardial infarction within 6 months prior to signing the ICF, New York Heart Association class III or IV, or clinically significant abnormalities of electrocardiogram (ECG) or cardiac function.
   3. History of coronary artery bypass graft surgery within 12 months prior to signing the ICF.
   4. History of severe liver function impairment as defined by Child-Pugh Class C, having an aspartate aminotransferase >3 × the upper limit of normal (ULN) or having an alanine aminotransferase >3 × ULN.
   5. History of severe kidney function impairment as defined by creatinine clearance (Cockcroft-Gault) <30 mL/min, being on dialysis, and/or having a serum creatinine >2 × ULN.
   6. History of known or suspected coagulopathy or uncontrolled anticoagulation (PLT count <100,000/μL; hemoglobin <12 g/dL; or hematocrit <35%).
   7. Loss of sensation in extremities or significant peripheral neuropathy.
6. As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
7. Has uncontrolled anxiety, psychiatric, or neurological disorder that, in the opinion of the Investigator, might interfere with study assessments.
8. Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
9. Has a known or suspected history of drug abuse over the last 6 months, a positive drug screen on the day of surgery, or a recent history of alcohol abuse over the last 6 months. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention-deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study at the discretion of the Sponsor.
10. Previously participated in a ZYNRELEF® or HTX-011 study.
11. Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half-lives (whichever is longer) prior to surgery, or is planning to take part in another clinical trial while participating in this study.
12. Has undergone 3 or more surgeries within 12 months prior to signing the Informed Consent Form, other than for diagnostic procedures (eg, colonoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-10-09 (Estimated); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Scores | 28 days
  Pain intensity scores using the NRS (either seated comfortably or lying down) on Day 0 before surgery, on arrival to the postanesthesia care unit(PACU), half hourly till departure from PACU, every 4 hours on the surgical floor until discharge on Postoperative Day 1 (POD1), then 48 hours,72 hours, Day 6 and Day 28.
Opioid rescue medication use | 28 days
  Date, time of administration, and amount of all opioid rescue medication taken through 72 hours in morphine equivalents. Data from discharge to 72 hours will be collected over a phone call. Subject daily diary to record if any opioids or acetaminophen were taken from 72 hours through Day 28.
Patient Global Assessment (PGA) | 28 days
  Patient Global Assessment (PGA) of pain control at 24, 48, and 72 hours, and on Day 28.
Discharge readiness assessment per the Modified Post Anesthetic Discharge Scoring System (MPADSS) | 24 hours
  Discharge readiness assessment per the Modified Post Anesthetic Discharge Scoring System (MPADSS) criteria at discharge on POD1
Subject's satisfaction with postoperative pain control | 6 days
  Subject's satisfaction with postoperative pain control at 24, 48, and 72 hours, and on Day 6 using a 5-point Likert scale.
Overall benefit of analgesia score (OBAS) | 28 days
  Overall benefit of analgesia score (OBAS) at 24, 48, and 72 hours, and on Day 28.
Time to Resume Exercise | 28 days
  Time taken to resume exercise after discharge in days. Subjects will be encouraged to report the time they resumed exercise. They will be asked at each communication as per the protocol.

SECONDARY OUTCOMES:
Demographics with height, weight, and BMI calculation. | 1 day
ACE and PHQ scores | 1 day
Medication history | 1 day
AEs from the time of drug application at surgery through Day 28. | 28 days
Episodes of nausea/vomiting and need for antiemetics postoperatively. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Raftopoulos, MD, Principal Investigator — Holyoke Medical Center
Locations (1):
- Holyoke Medical Center, Holyoke, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected in this study, including data dictionaries, will not be available to other researchers after the end of the study to protect the privacy of the participant data. Data will be in a database in the hospital's private Bariatric Drive. In addition, this will be a password-protected file that can be accessed only by the Principal Investigator, Research Coordinator, and Research Assistant.